CLINICAL TRIAL: NCT02127801
Title: A Single Dose Study of the Efficacy, Safety, Tolerability, and Pharmacokinetics of REGN1908-1909 in Allergic Rhinitis Subjects Challenged Intranasally With Allergen Extract
Brief Title: Single Ascending-dose Study of the Efficacy, Safety, Tolerability, and Pharmacokinetics of REGN1908-1909 in Allergic, Adult Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: R1908-1909-ALG-1325; U1111-1155-2258 (Other: World Health Organization); 2013-004950-68 (EudraCT Number)
Record Dates: First submitted 2014-04-29; First posted 2014-05-01 (Estimated); Last update posted 2020-12-16 (Actual); Status verified 2020-12

CONDITIONS: Allergy
MeSH Terms: conditions — Hypersensitivity

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | US Export: Yes

ARMS (2):
- Group A (Experimental): Participants in group A will receive REGN1908-1909
  Interventions: Drug: REGN1908-1909
- Group B (Experimental): Participants in group B will receive placebo
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: REGN1908-1909
  Arms: Group A
Drug: placebo
  Arms: Group B

SUMMARY:
The purposes of this study are to assess the efficacy, safety and tolerability of a single dose of REGN1908-1909 in allergic adult participants, to collect information about how much REGN1908-1909 is in blood over time and to collect information about how the body reacts to REGN1908-1909.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy men and women between the ages of 18 and 55
2. Positive allergen skin prick test
3. Willing and able to comply with clinic visits and study-related procedures
4. Provide signed informed consent

Exclusion Criteria:

1. Persistent, chronic, or active recurring infection requiring treatment with antibiotics, antivirals, or antifungals within 4 weeks prior to the screening visit
2. Any clinically significant (determined at the investigator's discretion) abnormalities observed during the screening physical examination
3. Onset of a new exercise routine or major change to a previous exercise routine within 4 weeks prior to the screening visit. Patients must be willing to maintain a similar level of exercise for the duration of the study and to refrain from unusually strenuous exercise for the duration of the trial
4. Hospitalization for any reason within 60 days prior to the screening visit
5. Participation in any clinical research study evaluating another investigational drug or therapy within 30 days or at least 5 half-lives (whichever is longer) of the investigational drug prior to the screening visit
6. Any medical or psychiatric condition that in the opinion of the investigator or Regeneron, would place the patient at risk, interfere with participation in the study or interfere with the interpretation of study results

The information listed above is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial and not all inclusion/ exclusion criteria are listed.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 74 (Actual)
Dates: Start 2014-10-31 (Actual); Primary Completion 2015-12-31 (Actual); Study Completion 2015-12-31 (Actual)

PRIMARY OUTCOMES:
Change in allergic symptom scale score | At day 8
  The primary endpoint is the change in allergic symptom scale score at day 8

SECONDARY OUTCOMES:
Incidence rate of treatment-emergent adverse events (TEAEs) through day 85 in participants treated with REGN1908-1909 or placebo | day 1 to day 85
Pharmacokinetic (PK) parameters of REGN1908- REGN1909 administration (i.e. how much REGN1908-1909 is in blood over time and how the body reacts to REGN1908-1909) | day 1 to day 85

CONTACTS AND LOCATIONS:
Locations (5):
- Groningen, Netherlands
- New Zealand (2):
  - Auckland
  - Christchurch
- Lund, Sweden
- London, United Kingdom

REFERENCES:
- [Derived] Shamji MH, Singh I, Layhadi JA, Ito C, Karamani A, Kouser L, Sharif H, Tang J, Handijiev S, Parkin RV, Durham SR, Kostic A, Orengo JM, DeVeaux M, Kamal M, Stahl N, Yancopoulos GD, Wang CQ, Radin AR. Passive Prophylactic Administration with a Single Dose of Anti-Fel d 1 Monoclonal Antibodies REGN1908-1909 in Cat Allergen-induced Allergic Rhinitis: A Randomized, Double-Blind, Placebo-controlled Clinical Trial. Am J Respir Crit Care Med. 2021 Jul 1;204(1):23-33. doi: 10.1164/rccm.202011-4107OC. PMID 33651675